CLINICAL TRIAL: NCT01594645
Title: The Impact of Selecting Acrosome Reacted Spermatozoa for ICSI- a Prospective RCT
Brief Title: The Clinical Impact of Selecting Acrosome Reacted Spermatozoa for ICSI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI moved from Hadassah
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013612- HMO-CTIL
Record Dates: First submitted 2012-05-03; First posted 2012-05-09 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2012-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Microscopy, Polarization; Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spermatozoa election using a polscope (Experimental): AR+ spermatozoa are selected for ICSI using a polscope
  Interventions: Procedure: Sperm selection by conventional / polarized light microscopy
- Control (Active Comparator): Spermatozoa for ICSI are selected based on morphology and motion under conventional light microscopy
  Interventions: Procedure: Sperm selection by conventional / polarized light microscopy

INTERVENTIONS:
Procedure: Sperm selection by conventional / polarized light microscopy — Selecting spermatozoa for ICSI using conventional and polarized light microscopy
  Other Names: Sperm selection, ICSI, polarized light

SUMMARY:
Presently spermatozoa for ICSI are selected based on morphology and motion, without determining if acrosome reaction (AR) had occurred during sperm preparation or not. Although not critical if the sperm is injected into the ooplasm, the occurrence of AR might might be an indicator of better spermatozoon quality and implantation potential, especially in severe OTA cases. It is impossible with conventional plain optic microscopy used in IVF units to determine in vivo (without fixation) if AR has occurred, and as a result spermatozoa are injected randomly. It is readily possible to distinguish AR+ from AR- spermatozoa using polarized light microscopy due to different bifriengance.

In this study the investigators seek to determine, by a prospective RCT, if selecting only acrosome reacted spermatozoa, in severe OTA cases, will improve the outcome of ICSI and the entire IVF process.

DETAILED DESCRIPTION:
A prospective RCT to determine the effect of polscope based spermatozoa selection for ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Female: normal uterine cavity and ovarian reserve. Male: TMC < 1000000 cells.

Exclusion Criteria:

* Female: Abnormal uterine anatomy, low ovarian reserve, contributing egg factor, PGD.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
fertilization rate | 24-72 h
  Determine the impact of AR+ spermatozoa selection of fertilization and in vitro embryonic development.

SECONDARY OUTCOMES:
Clinical pregnancy | up to 6 weeks
  The occurrence of clinical pregnancies in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Shufaro, MD PhD, Principal Investigator — HMO
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel